CLINICAL TRIAL: NCT02963129
Title: Treatment of Nasal Staphylococcus Aureus Colonization in Patients With Hereditary Hemorrhagic Telangiectasia With Recurrent Epistaxis.
Brief Title: Treatment of Nasal Staphylococcus Aureus Colonization in Patients With HHT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2666
Record Dates: First submitted 2016-08-09; First posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; Epistaxis
Keywords: Hereditary Hemorrhagic Telangiectasia; Epistaxis
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis | interventions — Mupirocin; Ointments

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mupirocina (Experimental): topical mupirocin nasal ointment and nasal solid petroleum jelly for 5 consecutive days and then just nasal solid petroleum jelly to complete the 60 total days
  Interventions: Drug: Mupirocin
- Control (Placebo Comparator): topical placebo nasal ointment and nasal solid petroleum jelly for 5 consecutive days and then just nasal solid petroleum jelly to complete the 60 total days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mupirocin — Mupirocin ointment in the nose for 5 days
  Other Names: Mupirocina 2% ointment
  Arms: Mupirocina
Other: Placebo — Placebo ointment in the nose for 5 days
  Other Names: ointment
  Arms: Control

SUMMARY:
Compare the frequency of epistaxis and quality of life related to nasal bleeding in patients with HHT colonized with sataphylococo before and after being treated with mupirocin ointment.

DETAILED DESCRIPTION:
Hereditary hemorrhagic telangiectasia is a vascular dysplasia characterized by the development of mucocutaneous telangiectasia and arteriovenous malformations in organs such as brain, lung, liver and tube digestivo. Is considered a rare disease, although It means that there is a substantial underdiagnosis. The overall prevalence is 1/5000.

Approximately 60% of the general population hosts strains of Staphylococcus aureus (S. aureus) intermittently and are called intermittent carriers, 20% represent persistent carriers harboring the same strain of S. aureus and 20% of the population are never carriers.

On this concept, one might think that HHT patients in whom there is an active and pathological vascular remodeling that causes bleeding, and inflammation is a known activator of abnormal angiogenesis; reducing an inflammatory factor as microbial through the eradication of nasal S. aureus could be useful to reduce bleeding in this population, directly impacting on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years with possible or confirmed HHT as diagnostic criteria Curaçao.
* Patients with nasal S. aureus colonization culture positive

Exclusion Criteria:

* Refusal to participate in the study or the informed consent process.
* Hypersensitivity or contraindication for topical mupirocin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Nosebleed by sadick scale | 60 days

SECONDARY OUTCOMES:
Prevalence of nasal colonization with Staphylococcus in patients with HHT by nasal cultive | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo MS Serra, MD, Principal Investigator — Staff of the Department of Clinical Medicine
Locations (2):
- Argentina (2):
  - Hospital Italiano de Buenos Aires, Peron 4190, Buenos Aires, Buenos Aires F.D.
  - Hospital Italiano de Buenos Aires, Gascon 450, Buenos Aires

IPD SHARING:
Plan to Share IPD: No